CLINICAL TRIAL: NCT06894771
Title: A Phase 1 Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-4700 as Monotherapy and in Combination With Pembrolizumab in Participants With Advanced or Metastatic Solid Tumors
Brief Title: A Study of MK-4700 Alone or With Pembrolizumab in Participants With Advanced or Metastatic Solid Tumors (MK-4700-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4700-001; MK-4700-001 (Other: MSD)
Record Dates: First submitted 2025-03-03; First posted 2025-03-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Malignant Neoplasm
Keywords: Head and Neck Squamous Cell Carcinoma; Melanoma; Non-small Cell Lung Cancer; Cervical Cancer; Triple Negative Breast Cancer; Urothelial Carcinoma; Renal Cell Carcinoma
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Transitional Cell; Carcinoma, Renal Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: MK-4700 (Experimental): Participants receive escalating doses every three weeks (Q3W) of MK-4700 for a maximum of 35 cycles (approximately 2 years; cycles are 21 days in length). Eligible participants enrolled in Arm 1 who experience progressive disease (PD) may cross over to Arm 2 to receive MK-4700 and pembrolizumab combination therapy.
  Interventions: Biological: MK-4700
- Arm 2: MK-4700 + Pembrolizumab (Experimental): Participants will receive MK-4700 and pembrolizumab Q3W for up to 35 cycles (approximately 2 years) or until PD, death, toxicity, or withdrawal of consent.
  Interventions: Biological: MK-4700; Biological: Pembrolizumab

INTERVENTIONS:
Biological: MK-4700 — Administered via subcutaneous (SC) injection
Biological: Pembrolizumab — Administered via intravenous infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm 2: MK-4700 + Pembrolizumab

SUMMARY:
The goal of this study is to learn about the safety of different doses of MK-4700 and if people tolerate them. The study will also measure what happens in a person's body over time when MK-4700 is given alone or with pembrolizumab (MK-3475) in order to find a dose that is safe, tolerated, and may work to treat certain types of cancer.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report who have experienced disease progression on or after prior anti-cancer treatments, or been intolerant to, or refused all treatment known to confer clinical benefit
* Has head and neck squamous cell carcinoma (HNSCC), melanoma (cutaneous), non-small cell lung cancer (NSCLC), cervical cancer, triple negative breast cancer (TNBC), urothelial carcinoma (UC), or renal cell carcinoma (RCC; clear cell, papillary)
* If human immunodeficiency virus (HIV) infected, must have well controlled HIV on antiretroviral therapy (ART)
* Has normal cardiac function

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* If HIV-infected with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease
* Has known additional malignancy that is progressing or has required active treatment within the past 2 years
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has active autoimmune disease that has required systemic treatment in the past 2 years except replacement therapy
* Has history of (noninfectious) pneumonitis/interstitial lung disease that required steroids
* Has current pneumonitis/interstitial lung disease
* Has active infection requiring systemic therapy
* Has known history of Hepatitis B (defined as Hepatitis B surface antigen reactive) or known active Hepatitis C virus infection
* Has had an allogeneic tissue/solid organ transplant in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | Cycle 1 (up to 21 days)
  The occurrence of any of the following toxicities during Cycle 1 will be considered a DLT, if assessed by the investigator related to study intervention administration:
  * Grade 4 nonhematologic toxicity
  * Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia
  * Any nonhematologic AE ≥Grade 3 in severity, with exceptions
  * Any Grade 3 or Grade 4 nonhematologic laboratory value, as with pre-specified exceptions
  * Any Grade 3 or Grade 4 laboratory abnormalities, with the exceptions
  * Febrile neutropenia Grade 3 or Grade 4
  * Prolonged delay (>2 weeks) in initiating Cycle 2 due to intervention-related toxicity
  * Any study drug toxicity that causes the participant to discontinue study drug during Cycle 1
  * Missing >25% of MK-4700 doses as a result of drug-related AEs during the first cycle
  * Grade 5 toxicity
Percentage of Participants Who Experience an Adverse Event (AE) | Up to approximately 4.5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants who Discontinue Study Treatment Due to an AE | Up to approximately 4.5 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve of MK-4700 | Predose and at prespecified time points during Cycles 1, 2, 3, 4, 5, 6, 7, and 10 up to approximately 7 months (Cycle length is 21 days)
  AUC is defined as the area under the concentration versus time curve. Blood samples will be collected at pre-specified timepoints to determine AUC.
Maximum Plasma Concentration (Cmax) of MK-4700 | Predose and at prespecified time points during Cycles 1, 2, 3, 4, 5, 6, 7, and 10 up to approximately 7 months (Cycle length is 21 days)
  Cmax is defined as the maximum concentration of MK-4700 observed in plasma after its administration and just prior to administration of the next dose. Blood samples will be collected at pre-specified timepoints to determine Cmax.
Minimum Plasma Concentration (Cmin) of MK-4700 | Predose and at prespecified time points during Cycles 1, 2, 3, 4, 5, 6, 7, and 10 up to approximately 7 months (Cycle length is 21 days)
  Cmin is defined as the minimum concentration of MK-4700 observed in plasma after its administration and just prior to administration of the next dose. Blood samples will be collected at pre-specified timepoints to determine Cmin.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- United States (2):
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0301), Hackensack, New Jersey
  - NEXT Oncology ( Site 0300), San Antonio, Texas
- Canada (2):
  - Princess Margaret Cancer Center ( Site 0101), Toronto, Ontario
  - Centre intégré de cancérologie du CHU de Québec Université Laval, Hôpital de l'Enfant-Jésus ( Site 0102), Québec, Quebec
- Israel (3):
  - Rambam Health Care Campus ( Site 0201), Haifa
  - Rabin Medical Center ( Site 0202), Petah Tikva
  - Sheba Medical Center ( Site 0200), Ramat Gan

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/